CLINICAL TRIAL: NCT06039059
Title: Influence of Risk Factors Such as Serum Cholesterol Level on ISR and Nonintervened Coronary Lesions
Brief Title: Influence of Risk Factors on ISR and Nonintervened Lesions
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Rf on ISR and nonintervented
Record Dates: First submitted 2023-09-07; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease; Multi Vessel Coronary Artery Disease
Keywords: ISR, nonintervened coronary lesions, risk factor
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Receiving PCI with nonintervened coronary lesion: Patients who received PCI with nonintervened coronary lesion.

SUMMARY:
This study enrolled patients who used to received PCI therapy with nonintervened coronary lesions. Baseline characteristics and laboratory testing were collected to find out the risk factor difference between ISR and nonintervened coronary lesions.

ELIGIBILITY:
Inclusion Criteria:

* (1) PCI therapy with drug-coated stents was performed in the past, and nonintervened coronary lesion remained except in the target vessel.

  (2) CAG was performed again due to re-examination, recurrent angina symptoms, positive treadmill exercise test or coronary CTA showing moderate to severe vessel diameter stenosis.

  (3) Long-term regular oral administration of statins and lipid monitoring were conducted after PCI.

Exclusion Criteria:

* Patients with a history of CABG, renal replacement therapy, autoimmune disease, and malignancy

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with multivessel lesions that had treated part of the vessels.
Sampling Method: Non-Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
LDL-C, mmol/L | Blood samples were collected after a 12-hour fast before CAG.
  Low-density cholesterol (LDL-C) is the cholesterol in low-density lipoprotein (LDL), which reflects how much LDL is present.

SECONDARY OUTCOMES:
HbA1c, % | Blood samples were collected after a 12-hour fast before CAG.
  Hemoglobin a1c (HbA1c) is the combination of hemoglobin and blood sugar. Its concentration in the blood is stable and is not affected by short-term blood sugar concentrations. Hemoglobin A1C has obvious clinical value in the diagnosis of diabetes.
ALT, U/L | Blood samples were collected after a 12-hour fast before CAG.
  Alanine aminotransferase (ALT) mainly exists in the plasma of liver cells, and the intracellular concentration is 1000-3000 times higher than that in serum. As long as 1% of liver cells are destroyed, it can double the serum enzyme. Therefore, alanine transaminase is recommended by the World Health Organization as the most sensitive detection index of liver function damage.
Scr, mmol/L | Blood samples were collected after a 12-hour fast before CAG.
  Serum creatinine (Scr) is a compound produced in muscles during the production of energy. Healthy kidneys filter creatinine from the blood. Creatinine is excreted in the urine as a metabolite and is a common measure of the kidney's filtration function. Creatinine this indicator belongs to the blood biochemical test, the higher the creatinine level, usually indicates the worse the kidney function.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tsao CW, Aday AW, Almarzooq ZI, Alonso A, Beaton AZ, Bittencourt MS, Boehme AK, Buxton AE, Carson AP, Commodore-Mensah Y, Elkind MSV, Evenson KR, Eze-Nliam C, Ferguson JF, Generoso G, Ho JE, Kalani R, Khan SS, Kissela BM, Knutson KL, Levine DA, Lewis TT, Liu J, Loop MS, Ma J, Mussolino ME, Navaneethan SD, Perak AM, Poudel R, Rezk-Hanna M, Roth GA, Schroeder EB, Shah SH, Thacker EL, VanWagner LB, Virani SS, Voecks JH, Wang NY, Yaffe K, Martin SS. Heart Disease and Stroke Statistics-2022 Update: A Report From the American Heart Association. Circulation. 2022 Feb 22;145(8):e153-e639. doi: 10.1161/CIR.0000000000001052. Epub 2022 Jan 26. PMID 35078371
- [Background] Patil CV, Nikolsky E, Boulos M, Grenadier E, Beyar R. Multivessel coronary artery disease: current revascularization strategies. Eur Heart J. 2001 Jul;22(14):1183-97. doi: 10.1053/euhj.2000.2497. No abstract available. PMID 11440491
- [Background] Rigattieri S, Biondi-Zoccai G, Silvestri P, Di Russo C, Musto C, Ferraiuolo G, Loschiavo P. Management of multivessel coronary disease after ST elevation myocardial infarction treated by primary angioplasty. J Interv Cardiol. 2008 Feb;21(1):1-7. doi: 10.1111/j.1540-8183.2007.00317.x. Epub 2007 Dec 12. PMID 18086133
- [Background] Nicolais C, Lakhter V, Virk HUH, Sardar P, Bavishi C, O'Murchu B, Chatterjee S. Therapeutic Options for In-Stent Restenosis. Curr Cardiol Rep. 2018 Feb 12;20(2):7. doi: 10.1007/s11886-018-0952-4. PMID 29435779
- [Background] Erdogan E, Bajaj R, Lansky A, Mathur A, Baumbach A, Bourantas CV. Intravascular Imaging for Guiding In-Stent Restenosis and Stent Thrombosis Therapy. J Am Heart Assoc. 2022 Nov 15;11(22):e026492. doi: 10.1161/JAHA.122.026492. Epub 2022 Nov 3. PMID 36326067
- [Background] Schupke S, Tiroch K. Acute Coronary Syndromes and the Nontarget Lesion. J Am Coll Cardiol. 2020 Mar 17;75(10):1107-1110. doi: 10.1016/j.jacc.2020.01.027. No abstract available. PMID 32164883
- [Background] Fukushima T, Yonetsu T, Aoyama N, Tashiro A, Niida T, Shiheido-Watanabe Y, Maejima Y, Isobe M, Iwata T, Sasano T. Effect of Periodontal Disease on Long-Term Outcomes After Percutaneous Coronary Intervention for De Novo Coronary Lesions in Non-Smokers. Circ J. 2022 Apr 25;86(5):811-818. doi: 10.1253/circj.CJ-21-0720. Epub 2021 Nov 18. PMID 34789614
- [Background] Kimura T, Morimoto T, Nakagawa Y, Kawai K, Miyazaki S, Muramatsu T, Shiode N, Namura M, Sone T, Oshima S, Nishikawa H, Hiasa Y, Hayashi Y, Nobuyoshi M, Mitudo K; j-Cypher Registry Investigators. Very late stent thrombosis and late target lesion revascularization after sirolimus-eluting stent implantation: five-year outcome of the j-Cypher Registry. Circulation. 2012 Jan 31;125(4):584-91. doi: 10.1161/CIRCULATIONAHA.111.046599. Epub 2011 Dec 27. PMID 22203694
- [Background] Glaser R, Selzer F, Faxon DP, Laskey WK, Cohen HA, Slater J, Detre KM, Wilensky RL. Clinical progression of incidental, asymptomatic lesions discovered during culprit vessel coronary intervention. Circulation. 2005 Jan 18;111(2):143-9. doi: 10.1161/01.CIR.0000150335.01285.12. Epub 2004 Dec 27. PMID 15623544
- [Background] Park MW, Seung KB, Kim PJ, Park HJ, Yoon SG, Baek JY, Koh YS, Jung HO, Chang K, Kim HY, Baek SH. Long-term percutaneous coronary intervention rates and associated independent predictors for progression of nonintervened nonculprit coronary lesions. Am J Cardiol. 2009 Sep 1;104(5):648-52. doi: 10.1016/j.amjcard.2009.04.052. PMID 19699339
- [Background] Kaneko H, Yajima J, Oikawa Y, Tanaka S, Fukamachi D, Suzuki S, Sagara K, Otsuka T, Matsuno S, Kano H, Uejima T, Koike A, Nagashima K, Kirigaya H, Sawada H, Aizawa T, Yamashita T. Long-term incidence and prognostic factors of the progression of new coronary lesions in Japanese coronary artery disease patients after percutaneous coronary intervention. Heart Vessels. 2014 Jul;29(4):437-42. doi: 10.1007/s00380-013-0382-6. Epub 2013 Jun 27. PMID 23807613